CLINICAL TRIAL: NCT06057831
Title: 18FDG-PET/MRI Imaging in Predicting Pathological Response to Total Neo-adjuvant Therapy in Rectal Cancer
Brief Title: PET/MRI in Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0034
Record Dates: First submitted 2023-08-18; First posted 2023-09-28 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All patients receive total neo-adjuvant therapy (TNT), depending on institutional policy
  Interventions: Radiation: Total Neo-adjuvant Therapy; Other: 18FDG-PET/MRI scan

INTERVENTIONS:
Radiation: Total Neo-adjuvant Therapy — * TNT incorporates chemotherapy with concurrent chemoradiotherapy (CRT) in any order.
  * Radiotherapy includes 5000 cGy/25 fractions over 5 weeks.
  * Chemotherapy regimen for Concurrent CRT: Capecitabine
  * Chemotherapy regimens used with TNT are: FOLFIRINOX x 6 cycles, 8-9 courses FOLFOX or 5-6 courses of CAPEOX delivered over 4-6 months.
  * The chemotherapy regimen or the order of treatment will be decided at the discretion of the patient's medical oncologist
Other: 18FDG-PET/MRI scan — 18FDG-PET/MRI scan within 4 weeks of commencing chemo-radiation and within 1 - 2 weeks before radical rectal cancer surgery.

SUMMARY:
The purpose of this study is to see which participants have a better treatment response using PET/MRI imaging to study the removed tumor, after they have received a total neoadjuvant therapy (TNT). The treatment choice of long course chemo-radiotherapy treatment will be determined by institutional policy.

The researchers will also be looking at whether this study could significantly improve the future management and quality of life of rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven adenocarcinoma of the rectum.
2. Clinical stage 2-3 rectal adenocarcinoma, cT3/4N0/M0 or Tx N1-2/M0, within 16 cm from anal verge (lesion below the sacral promontory).
3. Patients deemed suitable to undergo TNT followed by surgical resection.
4. Male or female ≥ 18 years of age.
5. ECOG/Zubrod status 0-2.
6. Able and willing to follow instructions and comply with the protocol.
7. Provide written informed consent prior to participation in the study.
8. Women of childbearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening if there is concern about pregnancy. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal.
9. If female of child-bearing potential and outside of the window of 10 days since the first day of the last menstrual period, concerned about pregnancy are not eligible for the study.
10. Females must not be breastfeeding (during treatment and at least 6 months from the last dose).
11. Male patients should agree that not donate sperm during the study (during treatment and at least 6 months from the last dose).
12. Patients of childbearing/reproductive potential should use highly effective birth control methods if indicated, as defined by the investigator, up to the period of finishing adjuvant chemotherapy. A highly effective method of birth control is defined as those that result in low failure rate (i.e., less than 1% per year) when used consistently and correctly.

Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.

Exclusion Criteria:

1. Patient receiving short course radiotherapy alone for rectal cancer.
2. Patient receiving standard TNT.
3. Patients with metastatic disease.
4. Prior pelvic radiotherapy or chemotherapy.
5. Patients in whom MRI is contra-indicated as per prevailing institutional guidelines (e.g. pacemakers, aneurysm clips, cochlear implant, implanted cardiac defibrillator).
6. Prior or concurrent malignancy (except non-melanomatous skin cancer) unless disease-free for at least 5 years.
7. Inability to lay in supine position for approximately one hour.
8. Nursing or pregnant females.
9. Age <18 years.
10. Previous and concurrent, experimental, chemotherapy, or radiotherapy treatment for primary rectal carcinoma.
11. Patients with malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease significantly affecting gastrointestinal (GI) function.
12. Patients with a known history of documented upper GI bleeding or upper GI ulcerative disease.
13. Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction.
14. Known current alcohol abuse.
15. Patients with symptomatic inflammatory bowel disease.
16. Patients with uncontrolled hypothyroidism.
17. Patients with chronic liver disease.
18. Patients known to be suffering from infection with HIV, Tuberculosis, Hepatitis C or Hepatitis B.
19. Any contra-indications for intravenous contrast.
20. History of anaphylactic reaction to medications or drug allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is pathological response (pCR) prediction with PET/MRI. | Week 29 - Week 31
  A 3-point scale will be used on PET/MRI assessment. When PET and MRI are concordant, the score remains unchanged. When MRI or PET are discordant, but one modality is definitive for complete response (e.g., MRI showing low intensity crescent at site of tumor or no uptake is identified on corresponding location on PET), a tumor regression grade (TRG) score of 1 will be assigned.
Correlation between PET/MRI reported pCR and complete(pCR) or incomplete response(non-pCR) to total neoadjuvant therapy determined by final pathology will be defined. | Week 31
  The pathologic response to the total neo-adjuvant therapy will be assessed generally using classification of tumor regression grade (TRG) defined by Mandard et al.

SECONDARY OUTCOMES:
To evaluate the significance of PET/MRI compared to MRI to predict response to TNT. | Week 29 - Week 31 (1 - 2 weeks before surgery)
  MRI imaging performed before and after TNT and the post TNT scans will be compared to baseline to identify the degree of regression. This comparison to baseline imaging will be performed to avoid misinterpretation of pseudotumor (inflammatory changes within normal rectal wall adjacent to regressed tumor) as residual tumor.
A feasibility study done to evaluate the benefit of using PET/MRI with respect to improved identification of the target and hence target delineation | Week 29 - Week 31 (1 - 2 weeks before surgery)
  Therapy plans are generated using image measures derived from standard radiotherapy plans or PET/MRI imaging. CT imaging is the standard imaging procedure used for radiotherapy treatment planning. In this clinical trial, a therapy plan will be generated from the initial PET/MRI imaging performed in the radiotherapy treatment position. This therapy plan will be compared with standard radiotherapy plans to evaluate the significance of using PET/MRI in radiotherapy treatment planning.

CONTACTS AND LOCATIONS:
Overall Officials: Kurian Joseph, Principal Investigator — AHS-CCI